CLINICAL TRIAL: NCT00469612
Title: Evaluating the Efficacy of NeuroVisions's NVC Treatment for Low Myopia
Brief Title: Evaluating NeuroVision's Neural Vision Correction (NVC) Myopia Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to lack of resources on part of investigators.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Donald Mutti, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006H0045
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Myopia
Keywords: Myopia; NeuroVision; Visual acuity; Contrast sensitivity
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): NeuroVision's NVC treatment for low myopia
  Interventions: Device: NeuroVision's NVC treatment for Low Myopia
- B (No Intervention): The subjects in this group will serve as controls and will be the no intervention group.

INTERVENTIONS:
Device: NeuroVision's NVC treatment for Low Myopia — NeuroVision's NVC vision correction technology is a method in the treatment of low myopia as the technology is directed at specific neuronal interactions at the level of the visual cortex (area responsible for vision in the brain).
  The subject will be exposed to a set of visual stimulations (pattern with black and white lines) and visual threshold level will be obtained. The subject will look at these patterns on a computer. The treatment will be applied in successive 30-40 minute sessions, administered 2-3 times a week, for a total of 40 sessions. Every 5 sessions, subject's visual performance (visual acuity and CSF) will be tested in order to continuously monitor a subject's progress.
  Arms: A

SUMMARY:
The purpose of the present study is to carry out a trial to evaluate the clinical efficacy of the NeuroVision Low Myopia Treatment.

The specific questions to be answered are:

1. Is there an improvement in vision following the treatment without bringing about a change in the subject's prescription for glasses?
2. Can any treatment effect be seen at 6 months and 12 months after the termination of the treatment?

DETAILED DESCRIPTION:
Myopia and its treatment modalities are one of the widely studied areas in vision research. So far all the treatment options have been optical i.e., patients with myopia are either corrected with spectacles, contact lenses or refractive surgery to provide clear vision. NeuroVision's NVC vision correction technology will be a novel method in the treatment of low myopia as the technology is directed at specific neuronal interactions at the level of the visual cortex (area responsible for vision in the brain). It uses a non-invasive, patient-specific treatment that purports to improve neuronal efficiency and induce improvement in the overall ability to see due to a reduction in noise and increase in signal strength. As visual perception quality depends both on the input received through the eye and the processing in the visual cortex, NeuroVision's technology is hypothesized to compensate for blurred (myopic) inputs, by enhancing neural processing.

We will conduct a clinical evaluation of the effectiveness of this system. The subject will be exposed to a set of visual stimulations (pattern with black and white lines) and visual threshold level will be obtained. The subject will look at these patterns on a computer. The treatment will be applied in successive 30-40 minute sessions, administered 2-3 times a week, for a total of 40 sessions. Every 5 sessions, subject's visual performance (visual acuity, ability to see letters of varying size, and CSF, ability to see black and white lines of varying contrast) will be tested in order to continuously monitor a subject's progress. At the end of a session, the data will be sent to the NeuroVision Web Server. Proprietary algorithmic software will analyze the patient's performance and progress and will generate the parameters for the next treatment session. The purpose of the study is to assess the effect on corrected or uncorrected visual performance following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age should be between 18 to 59 years
* Spherical equivalent in the worst eye should not exceed -1.5 DS and the astigmatism should not exceed -0.75 DC.
* The subject's refractive status is stable, with no increase beyond 0.5D in sphere or cylinder over the last six months. That is, the subject's spectacle prescription should not differ from the auto-refraction value by 0.50D.
* Unaided visual acuity is 0.6 LogMAR or better in the eye with the poorer unaided acuity
* Unaided visual acuity is 0.1 LogMAR or worse in the eye with better unaided acuity
* Unaided visual acuity difference between both eyes is less than 0.3 LogMAR
* Best-corrected visual acuity is 0.04 LogMAR or better in both eyes.
* The subject should be aware that the study has the following features:

  1. The recommended pace for the treatment sessions is at least 3 sessions per week.
  2. Interruptions should not be longer than 2 weeks during the treatment course. Note: The subject is free to voluntarily withdraw from the study at any time.

Exclusion Criteria:

* The subject suffers from any other visually disabling eye disease(s) or other causes for the reduced visual acuity, aside from myopia and/or astigmatism
* The subject suffers from myopia-related visual complications resulting in visual loss, including myopic macular degeneration, myopic cataract and previous or pre-existing myopic retinal detachment.
* The subject is suffering from Diabetes Mellitus.
* The subject suffers from Migraines
* The subject suffers from Epilepsy
* The subject is pregnant. (It is not recommended to include pregnant women because of the expected visual fluctuations. The NV treatment , basically using a computer, has no impact on the pregnancy.) No pregnancy testing will be done but will be identified through verbal history. The study has use of tropicamide drug (dilation drops) and proparacaine (topical anesthetic), which are a routinely used eye drop in everyday clinical practice and no adverse effects have been reported so far on pregnant women or fetus.
* The subject has an activity limitation due to medical disorders (including migraines, seizure disorders, etc.), medications, or emotional status that might potentially impair the subject's ability to perform the treatment.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald O Mutti, OD, PhD, Principal Investigator — Ohio State University
Locations (1):
- College of Optometry, The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Polat U, Sagi D. The architecture of perceptual spatial interactions. Vision Res. 1994 Jan;34(1):73-8. doi: 10.1016/0042-6989(94)90258-5. PMID 8116270
- [Background] Polat U, Sagi D. Lateral interactions between spatial channels: suppression and facilitation revealed by lateral masking experiments. Vision Res. 1993 May;33(7):993-9. doi: 10.1016/0042-6989(93)90081-7. PMID 8506641
- [Background] Polat U, Sagi D. Spatial interactions in human vision: from near to far via experience-dependent cascades of connections. Proc Natl Acad Sci U S A. 1994 Feb 15;91(4):1206-9. doi: 10.1073/pnas.91.4.1206. PMID 8108388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two subjects were recruited when study began, but before data were collected the study was terminated due to lack of resources.
Groups:
- NeuroVision's NVC Treatment for Low Myopia: NeuroVision's NVC treatment for low myopia
  NeuroVision's NVC treatment for Low Myopia: NeuroVision's NVC vision correction technology is a method in the treatment of low myopia as the technology is directed at specific neuronal interactions at the level of the visual cortex (area responsible for vision in the brain).
  The subject will be exposed to a set of visual stimulations (pattern with black and white lines) and visual threshold level will be obtained. The subject will look at these patterns on a computer. The treatment will be applied in successive 30-40 minute sessions, administered 2-3 times a week, for a total of 40 sessions. Every 5 sessions, subject's visual performance (visual acuity and CSF) will be tested in order to continuously monitor a subject's progress.
- No Intervention Group: The subjects in this group will serve as controls and will be the no intervention group.
Period: Overall Study
Arm/Group | NeuroVision's NVC Treatment for Low Myopia | No Intervention Group
Started | 2 | 0
Completed | 0 (Subjects enrolled, but no data collected. Study terminated before data collection.) | 0
Not Completed | 2 | 0
Not completed — Study terminated before data collected | 2 | 0

BASELINE CHARACTERISTICS:
Population: Two subjects were enrolled, but no data were collected because study was terminated due to lack of resources.
Groups:
- Total: Total of all reporting groups
Arm/Group | NeuroVision's NVC Treatment for Low Myopia | No Intervention Group | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 0 |  | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Time Frame: Every 5th visit
Population: Two subjects were enrolled, but no data were collected because study was terminated due to lack of resources.
Arm/Group | NeuroVision's NVC Treatment for Low Myopia | No Intervention Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Contrast Sensitivity Function
Time Frame: Every 5th visit
Population: Two subjects were enrolled, but no data were collected because study was terminated due to lack of resources.
Arm/Group | NeuroVision's NVC Treatment for Low Myopia | No Intervention Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Refractive Error
Time Frame: Every 10th visit
Population: Two subjects were enrolled, but no data were collected because study was terminated due to lack of resources.
Arm/Group | NeuroVision's NVC Treatment for Low Myopia | No Intervention Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | NeuroVision's NVC Treatment for Low Myopia | No Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
Two subjects were enrolled, but no data were collected because study was terminated due to lack of resources.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes